CLINICAL TRIAL: NCT02369562
Title: A Retrospective Analysis of Failures/Complications With Oral Implants
Brief Title: A Retrospective Analysis of Failures of Oral Implants
Status: Completed | Type: Observational
Sponsor: Malmö University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Principal Investigator, Bruno Ramos Chrcanovic, DDS, MSc, PhD student, Malmö University
Other Study IDs: Dnr 2014/598
Record Dates: First submitted 2015-02-10; First posted 2015-02-24 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Dental Implant Failure; Periodontal Bone Loss
Keywords: Dental implants; Periodontal Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dental implant patients: All patients rehabilitated with dental implants.
  Interventions: Procedure: Evaluation of the failure rate of dental implants

INTERVENTIONS:
Procedure: Evaluation of the failure rate of dental implants — Evaluation of the failure rate of dental implants, from the time of implant insertion (any time between 1980 and August 31st 2014) until September 2015
  Other Names: Implant failure rate assessment

SUMMARY:
The purpose of this retrospective study is to investigate and identify factors associated with the failure of dental implants within the population rehabilitated with dental implants at the Folktandvården Specialistklinik in Malmö (Spårvägsgatan 12, 214 27, Malmö).

DETAILED DESCRIPTION:
This is a retrospective study that involves collecting information about the past and comparing that with contemporary information collected from the same cases. The patients' dental records' archive and the digital dental records of the Folktandvården Specialistklinik in Malmö will be scrutinized. The patients will be retraced in the Swedish Personal Data System and will be invited for a recall visit with a clinical and radiographic examination. The patients will then be informed of the design of the study through the reading of the Form for Patient Information and the Informed Consent in Swedish and verbally. In case the patient is not willing to pay a recall visit, only the data of the patient's records will be used, under the patients' approval.

The data from the patients' records will be directly inserted to a computer file of the statistical software Statistical Package for the Social Sciences (SPSS Inc., Chicago, USA). The additional follow-up information from the patients' recall visit will be collected in specific forms and then inserted to the previously mentioned computer file. All dental implants inserted will be included in the study. Data will be categorized as surgical, implant-specific, patient-related, anatomic, loading conditions, prosthetic, and trans- and postoperative complications.

Periapical radiographies of the patients' digital record will be neatly filed in a computer file. Periapical radiographies that could possibly exist in celluloid film will be digitalized. From each patient, additional radiographs will be selected from the patient's record, based on availability in several time intervals. At the recall consultation, new periapical radiographies will be taken. The reference point will be established at the implants-abutment junction, and the marginal bone level measurement will be performed by using the Image J software.

ELIGIBILITY:
Inclusion Criteria:

* All treated patients with dental implants placed and restored at the Avdelning för Oral Protetik at the Folktandvården Specialistklinik in Malmö with an available dental record;
* Patients having read, understood, and signed the Form for Patient Information and the Informed Consent.

Exclusion Criteria:

* Patients not willing to give their permission to scrutinize their records;
* Lack of enough data in the patients' dental records.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population rehabilitated with dental implants at/or referred to prosthetic rehabilitation at the Avdelning för Oral Protetik at the Folktandvården Specialistklinik in Malmö.
Sampling Method: Probability Sample
Enrollment: 2670 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Survival of implants | Including implants placed from 1980 until August 31st 2014
  Time from the surgical placement of implants until the last follow-up or until its failure

SECONDARY OUTCOMES:
Marginal bone loss | Including implants placed from 1980 until August 31st 2014
  Time from the surgical placement of implants until the last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bruno R Chrcanovic, DDS MSc, Principal Investigator — Malmö University; Ann Wennerberg, DDS PhD, Study Director — Malmö University; Tomas Albrektsson, MD PhD, Study Director — Göteborg University / Malmö University; Jenö Kisch, DDS, Study Chair — Region Skane
Locations (1):
- Folktandvården Specialistklinik, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chrcanovic BR, Kisch J, Albrektsson T, Wennerberg A. Factors Influencing Early Dental Implant Failures. J Dent Res. 2016 Aug;95(9):995-1002. doi: 10.1177/0022034516646098. Epub 2016 May 4. PMID 27146701